CLINICAL TRIAL: NCT03463720
Title: Outcome for Patients With War-Associated Extremity Wound Infection
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The International Federation of Red Cross and Red Crescent Societies (Other)
Responsible Party: Principal Investigator, Jonas Malmstedt, Principal Investigator, Karolinska Institutet
Other Study IDs: KISOS003
Record Dates: First submitted 2018-02-22; First posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Extremity wound: Patients with extremity wounds. Infected and not infected patients will be compared.
  Interventions: Other: Infected; Other: Not infected

INTERVENTIONS:
Other: Infected — Extremity wound, infected
Other: Not infected — Extremity wounds, non-infected

SUMMARY:
Extremity wounds and fractures constitute the majority of war-associated traumatic injuries, both for civilians and combatants. War-associated injuries are often contaminated with foreign material, leading to infection. Wound infections is considered a major risk to life and restoration of function in war-wounded patients surviving past the first hours. In a cohort study the investigators aim to assess whether the infection itself affects patient outcome (i.e. amputation, death) when comparing patients with and patients without infection.

DETAILED DESCRIPTION:
Armed violence has occurred intermittently in northwestern Pakistan and neighboring Afghanistan since the beginning of the 1980s. In 1981 the International Committee of the Red Cross (ICRC) opened a hospital in Peshawar, Pakistan, to care for the injured from the armed conflict in Afghanistan. In 2004 the number of patients increased as a result of the emerging divergence between the State of Pakistan and militant groups in the Northwestern Pakistan. Yearly about 1000 patients with war-associated injuries, predominantly caused by gunshots and explosive devices have been treated for free at the ICRC hospital in Peshawar. The hospital is now closed.

War-associated injuries are generally treated according to the ICRC war surgical protocol. Research on the epidemiology of and risk factors for wound infection in patients with war-associated injuries is limited and primarily include military combatants, leading to a selection of young males. Due to the use of body armor and forward surgical teams this data may not be applicable to a civilian setting. It is unknown to what extent wound infection itself is a factor contributing to serious complications such as amputation and death. Knowledge is needed to gear resources towards those most in need. This research makes use of a unique database that contains both civilians and combatants of both sexes and all ages. The investigators aim to assess whether the infection itself affects patient outcome (i.e. amputation, death) when comparing patients with and patients without infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients that have received treatment for war-associated extremity wounds
* Patients that present at the hospital within 72 hours of injury
* Patients with valid data on baseline wound status.

Exclusion Criteria:

• Patients that are re-admitted during the study period, i.e. patients that received treatment during the study period and are later re-admitted will only be counted as one patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients treated at the hospital in Peshawar between September 27, 2010 and May 9, 2012 that meet eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 843 (Actual)
Dates: Start 2010-09-27 (Actual); Primary Completion 2012-05-09 (Actual); Study Completion 2012-05-09 (Actual)

PRIMARY OUTCOMES:
Amputation | From hospital admission to discharge, an average of 15 days
  In-hospital extremity amputation. Upper or lower extremity, all levels.

SECONDARY OUTCOMES:
Death | From hospital admission to discharge, an average of 15 days
  In-hospital death

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Malmstedt, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- International Committee of the Red Cross hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No
The use of identification numbers will ensure anonymity of the data. All data will remain confidential throughout the data entry and analysis process by encryption. Individual patient data will not be distributed outside the study location, or appear in any report or publication.